CLINICAL TRIAL: NCT00137891
Title: Phase I Study Comparing Pharmacokinetics and Safety Profile of Thyrogen Versus a Modified Release of Recombinant Human Thyroid Stimulating Hormone
Brief Title: Study Comparing Thyrogen Versus a Modified Release of Recombinant Human Thyroid Stimulating Hormone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THYR01205
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Multinodular goiter

INTERVENTIONS:
Drug: Modified Release rhTSH

SUMMARY:
Forty-six (46) eligible, healthy subjects who provide written informed consent will be enrolled to participate in a 2 arm parallel group study to assess and compare the pharmacokinetics and safety profile of Thyrogen dosed at 0.1 mg versus a modified release formulation of recombinant human thyroid stimulating hormone (rhTSH) dosed at 0.1 mg. Ten (10) of these subjects will have the thyroid uptake of radioiodine (123I) measured at baseline and following their single dose of study medication. All doses will be administered via intramuscular (IM) injection.

Following confirmation of study eligibility, subjects will be randomized in a 1:1 ratio to receive either a single administration of 0.1 mg of Thyrogen (THYR) or 0.1 mg of the modified release.

Randomization will be stratified by whether or not patients will have the thyroid uptake of radioiodine (123I) measured following their single dose of study medication. Five (5) patients in each treatment arm will have uptake measured, while 18 in each arm will not.

Each subject will have blood samples taken to determine the pharmacokinetics of serum TSH at -12 hours and just prior to dosing and at various hours up to 14 days following the administration of Thyrogen or the modified release formulation. In addition, for the evaluation of pharmacodynamics, each subject will have samples of blood taken to determine serum free T4, total T4, free T3, and total T3 at -12 hours and just prior to dosing and at various hours up to 14 days following the administration of study treatments.

All subjects will undergo a 12-lead electrocardiogram (ECG) just prior to dose administration and 1, 2, 3, 4, 5, 7, 10 and 14 days following study treatment administration. In addition, subjects will undergo 24 hours of Holter monitoring at baseline and four (4) consecutive 24-hour Holter monitoring sessions post treatment to yield a total of 96 hours of continuous monitoring of cardiac function following treatment administration. All subjects will undergo ultrasound evaluations to determine thyroid volume at baseline and 48 hours following treatment administration.

Twenty-four hours following the administration of Thyrogen or the modified release formulation, a subset of five (5) subjects in each treatment arm will receive a dose of 123I prepared to be 400µCi on the day of radioiodine administration based on the utilized nuclear pharmacy's calibration schedule. Thyroid gland uptake will be measured via a probe in these 10 subjects at 6, 24 and 48 hours following radioiodine administration.

Blood chemistry, complete blood count (CBC), urinalysis and a physical exam will be conducted 14 days after treatment administration, or at the time of early termination, as a final safety assessment.

Each subject's duration of study participation will be approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Committed to follow the protocol requirements as evidenced by providing written informed consent prior to any study-related procedures being performed
* Males or females, in good general health, between the ages of 18 and 40, inclusive. Females of childbearing potential must be on a stable hormonal contraceptive regimen (defined as > 6 months continuous use) and/or utilize a double barrier method, i.e., condom and foam. It is recommended that female sexual partners of male subjects utilize the above described method of birth control while their partners are participating in the study.
* A negative serum pregnancy test prior to entering the study (all women regardless of child bearing potential)
* Physical examination, including vital signs and laboratory assessments that are within normal limits at the time of screening. If abnormalities are noted, they must be deemed clinically insignificant, based on the investigator's judgment, to satisfy inclusion criteria.
* Electrocardiogram (ECG) and Holter results within normal limits at screening. Subjects who have ECG findings of occasional premature atrial beats, abnormal PR intervals not associated with supraventricular tachycardia (SVT) or heart block, right bundle branch block, sinus tachycardia at rest (heart rate [HR] < 100 beats per minute [BPM]) and sinus bradycardia (HR > 50 BPM) may be included in this study.
* Urine and plasma drug screens are negative for drugs of abuse at the time of screening
* Willing and able to abstain from alcohol 48 hours prior to and post each administration of Thyrogen and otherwise limit all alcohol consumption to < 2 drinks per day while participating in the study
* Absence of or current smoking habit of < 10 cigarettes per day while participating in the study
* Baseline levels of total T3, free T3, free T4, T4, and TSH levels within the normal range
* Body mass index (BMI) < 30

Exclusion Criteria:

* Any history of cardiovascular disease
* Uncontrolled hypertension as defined by a resting blood pressure of > 140/90 mm Hg (resting defined as 5 minutes sitting/supine position)
* Currently or within the past 5 years a history of malignancy, other than squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix
* A concurrent major medical disorder (e.g., documented cardiac disease, debilitating cardiopulmonary disease, advanced renal failure, advanced liver disease, advanced pulmonary disease, or advanced cerebral vascular disorder) and may be too ill to adequately comply with the requirements of this study
* ECG or Holter abnormalities that may be suggestive of underlying cardiac disease including: left atrial abnormality and/or left ventricular hypertrophy, frequent ectopic or multifocal atrial beats, frequent premature ventricular beats, significant conduction abnormalities such as widened QRS, left bundle branch block, significant axis deviation, atrial fibrillation or flutter, frequent premature ventricular contractions or ventricular tachycardia (including torsades de point), repolarization changes suggestive of myocardial ischemia (e.g., ST-T wave abnormalities suggestive of ischemia), evidence of a previous myocardial infarction, atrioventricular (AV) nodal reentrant tachycardia or tachycardias associated with preexcitation/accessory pathway syndromes and high grade AV block
* A non-thyroidal condition known to affect 123I uptake (e.g., congestive heart failure class III or IV, renal failure)
* Currently taking drugs that may affect thyroid or renal function (e.g., corticosteroids, diuretics, lithium, amiodarone, or other prescribed iodine-containing medication)
* Women of childbearing potential unless taking medically acceptable contraceptive precautions
* Women who are pregnant or lactating
* A current diagnosis or recent history, within the past 2 years, of alcoholism, drug abuse, or severe emotional, behavioral or psychiatric problems that, in the opinion of the Investigator, would hinder adequate compliance with the requirements of this study
* Currently participating in another investigational drug study or have participated in such a study within 30 days of their enrollment in this study
* Have schedule or travel plans that prevent the completion of all required visits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46
Dates: Start 2005-06; Study Completion 2005-08

PRIMARY OUTCOMES:
To assess and compare the pharmacokinetics (PK) of a single intramuscular (IM) administration of 0.1 mg of Thyrogen versus a single IM administration of 0.1 mg modified release formulation of rhTSH in healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- SFBC International, Miami, Florida, United States